CLINICAL TRIAL: NCT00353535
Title: Phase 1 Study of TLI Pretransplant to Prevent Recurrence of FSGS in the Graft
Brief Title: Total Lymphoid Irradiation (TLI) to Prevent Focal Segmental Glomerulosclerosis (FSGS)Recurrence in the Renal Graft
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLIFSGSusp
Record Dates: First submitted 2006-07-17; First posted 2006-07-18 (Estimated); Last update posted 2006-07-18 (Estimated); Status verified 2005-09

CONDITIONS: Glomerulosclerosis, Focal
Keywords: glomerulosclerosis, focal; pretransplant immunosuppression; total lymphoid irradiation; renal transplant; recurrence
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental; Recurrence

INTERVENTIONS:
Procedure: Total Lymphoid irradiation

SUMMARY:
The purpose was study the immunosuppression using total lymphoid irradiation plus Csa, MMF and prednisone pretransplant to prevent focal segmental glomerulosclerosis recurrence in the renal graft

DETAILED DESCRIPTION:
Focal and segmental glomerulosclerosis (FSGS) is resistant to treatment with immunosuppressants and after transplant, 40% of such patients have recurrences in renal allograft. The purpose of this trial was to use Total Lymphoid Irradiation (TLI) plus mycophenolate mofetil (MMF), cyclosporine A (CsA) and prednisone (PRED) to prevent recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients (age > 18 years)
* Biopsy-proven primary FSGS
* End-stage renal failure at presentation or prior allograft loss due to recurrent FSGS.
* Signed the informed consent before entering in the study.

Exclusion Criteria:

* Age < or equal 18 years
* No biopsy-proven FSGS
* Without living donor to perform the transplant
* No signed the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2000-01; Study Completion 2002-12

PRIMARY OUTCOMES:
Efficacy of immunosuppression using TLI plus CsA, MMF and Pred in prevent recurrence of FSGS after the renal transplant

SECONDARY OUTCOMES:
Morbidity and mortality ot the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Chocair, Prof. PhD, Principal Investigator — Renal Transplant Unity - Hospital das Clinicas - Medicine School - University of Sao Paulo - Brazil; Rosangela Villar, MD, Principal Investigator — Assistent doctor and Medical Supervisor of Division of Radiotherapy - Institute of Radiology - Hospital das Clinicas - University of Sao Paulo
Locations (1):
- Hospital das Clinicas - Division of Urology and Radiotherapy - University of Sao Paulo, São Paulo, São Paulo, Brazil